CLINICAL TRIAL: NCT04173923
Title: Long Term Follow-up of Cervical Myelopathy Inpatients Treated With Integrated Complementary and Alternative Medicine
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2019-05
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cervical Myelopathy
Keywords: Cervical Myelopathy; Korean medicine treatment
MeSH Terms: interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine will be administered in water-based decoction (120ml) and dried powder (2g) form (Ostericum koreanum,Eucommia ulmoides, canthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, aposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycinemax, Atractylodes japonica) at the physician's discretion.
  Other Names: Traditional herbal medicine
Procedure: Chuna manual medicine — Chuna is a Korean manual therapy directed at the spine and joints that incorporates various spinal manual medicine techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manual medicine will be administered to the pelvic, lumbar, thoracic, and cervical vertebrae at the physician's discretion.
  Other Names: Chuna manipulation
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Hyeopcheok (Huatuo Jiaji, EX B2), Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea) at the physician's discretion.
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Procedure: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary regardless of type or dose, and patterns of use will be investigated and recorded as a pragmatic clinical study.

SUMMARY:
Model of this study is a combined both retrospective chart review and follow up survey. Data of 4 hospitals will be used to find out the efficacy of conservative treatment in cervical myelopathy.

DETAILED DESCRIPTION:
Cervical myelopathy is known as Its symptoms are progressively worsened, and there are only a small amount of positive outcomes other than surgery.

However, as with other spinal and nerve disorders, non-surgical treatments are getting more attention in terms of patient safety, and because they provide patients with more choice in treatment than in terms of surgical treatment, they can provide closer approach to patient-centered care.

Physical therapy and medication are well known for the currently known non-surgical and conservative treatments, but research reported on the treatment of cervical myelopathy by using Korean medicine treatment so far has its weak level. Therefore, it is expected that this study will demonstrate the efficacy of the treatment of cervical myelopathy in Korean medicine treatment and will further pave the way for non-surgical treatment of spinal myelopathy.

Therefore, The investigators conducted observational trial to analyze the effectiveness of Korean medicine treatment in spinal myelopathy. Retrospective data will be extracted using electronic medical records and computerized data of hospitalized patients. Based on this, investigators will conduct research in the form of prospective survey and analyze the causal relationship and factors using the two data.

The hospital's medical records will be used to analyze the patient's condition during the hospitalization period and to determine the situation after the end of treatment through questionnaire. The questionnaire will be developed after consultation with experts from musculoskeletal system and related societies, and will be used for the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been hospitalized with symptoms of neurological defects such as muscle weakness in the upper extremity or sensory abnormalities, or impaired walking due to weakness in the lower extremity at Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital and Incheon Jaseng Korean Medicine Hospital from Jan 2011 to Oct 2018.
* Patients diagnosed with 'Cervical myelopathy' finding and able to check the pressure and damage of the spinal cord (high signal shading) of the EMR imaging (T2-weighted MRI scan of C-spine)
* Patients who agreed voluntarily to participate in verbal consent

Exclusion Criteria:

* Patients whose chief complaint is not cervical myelopathy or who do not have the neurological defect of upper extremity or lower extremity
* If the cause of the neurological defect of the upper and lower extremities is not caused by the spine or tissue
* Patients who do not agree to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who ended up the hospitalization and treatment in Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, Incheon Jaseng Korean Medicine Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Cervical spinal surgery status after discharge | Finish survey by Jan 2020
  The investigators will survey whether the patients had surgery after discharging from 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Incheon Jaseng Korean Medicine Hospital.

SECONDARY OUTCOMES:
Cervical spinal surgery recommendations before hospitalization | Finish survey by Jan 2020
  The investigators will survey whether the patients were recommended before hospitalization in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Incheon Jaseng Korean Medicine Hospital).
Symptom reoccurrence experience lasting for more than a month after treatment is closed | Finish survey by Jan 2020
  The investigators will survey whether the patients experienced symptom reoccurrence lasting for more than a month after treatment is closed after hospitalization in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Incheon Jaseng Korean Medicine Hospital).
Whether symptoms that are uncomfortable in daily life exists | Finish survey by Jan 2020
  The investigators will survey whether the patients feel uncomfortable daily life symptoms after hospitalization in 4 hospitals(Haeundae Jaseng Korean Medicine Hospital, Jaseng Korean Medicine Hospital, Bucheon Jaseng Korean Medicine Hospital, and Incheon Jaseng Korean Medicine Hospital).
Whether currently being treated for neck or upper extremity symptoms | Finish survey by Jan 2020
  The investigators will survey whether the patients are currently being treated for neck or upper extremity symptoms
Numeric Rating Scale of Neck and upper extremity pain | Finish survey by Jan 2020
  The investigators will survey Numeric Rating Scale(NRS) scores of neck and upper extremity at the time of the disease and current symptoms.
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Neck Disability Index | Finish survey by Jan 2020
  The investigators will survey current Neck Disability Index (NDI) scores. NDI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
EuroQol 5-dimensions 5-levels | Finish survey by Jan 2020
  The investigators will survey current EuroQol 5-dimensions 5-levels scores. The EQ-5D-5L is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems).
Patient Global Impression of Change | Finish survey by Jan 2020
  The investigators will survey current Patient Global Impression of Change scores.
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Study Chair — Jaseng Medical Foundation
Locations (1):
- Haeundae Jaseng Hospital of Korean Medicine, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided